CLINICAL TRIAL: NCT04451265
Title: Diagnostic Accuracy of Optimized Diffusion-Weighted Imaging for Detecting Anterior Ischemic Optic Neuropathy
Acronym: DACODAC
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GPN_2020_6
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Neuro-Ophthalmology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRI — Diffusion sequence (8 minutes long) added to the initial MRI

SUMMARY:
The patient presents to the ophthalmological emergencies and / or to the internal medicine department. NOIA clinical discovery Patient referred in radiology for brain and visual MRI. The two sequences added by the research (8 minutes) will be added to that of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patient with suspected NOIA, evoked after clinical examination by a specialized ophthalmologist
* For which a brain and visual MRI is planned
* Express consent to participate in the study
* Affiliate or beneficiary of a Social Security scheme

Exclusion Criteria:

* Contraindication to MRI (electrical device, metallic foreign body, claustrophobia)
* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspected NOIA, discussed after clinical examination by a specialist ophthalmologist
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Study the sensitivity of the High resolution Diffusion sequence in the detection of NOIA, evaluated by a DWI hypersignal and an ADC hyposignal of the optic nerve | basline

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de LILLE, Lille, Lille
  - Fondation A De Rothschild, Paris, PARIS
  - Chu Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No